CLINICAL TRIAL: NCT07177482
Title: ImmunoPET Targeting Trophoblast Cell-surface Antigen 2 (Trop-2) in Craniopharyngioma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deling Li (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor-Investigator, Deling Li, Professor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BTHospital-N-010
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Craniopharyngioma
Keywords: Positron-Emission Tomography; Diagnosis
MeSH Terms: conditions — Craniopharyngioma; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-MY6349 PET/CT (Experimental): Each subject receives a single intravenous injection of 68Ga-MY6349 and undergoes PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 68Ga-MY6349 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-MY6349 PET/CT — Each subject receives a single intravenous injection of 68Ga-MY6349 and undergoes PET/CT imaging within the specified time.

SUMMARY:
This study aims to investigate 68Ga-MY6349, an immune-PET tracer targeting trophoblast cell surface antigen 2 (Trop2), for the noninvasive diagnosis of craniopharyngioma in vivo.

DETAILED DESCRIPTION:
The trophoblast cell surface antigen 2 (Trop2), encoded by the TACSTD2 gene, is a transmembrane glycoprotein that regulates epithelial malignant transformation and proliferation. Trop2 has been reported to be overexpressed in various epithelial tumors, including craniopharyngioma. 68Ga-MY6349, an immune-PET tracer targeting Trop2, has demonstrated high specificity and sensitivity in visualizing other Trop2-high solid tumors. In this research, patients with primary or recurrent craniopharyngioma scheduled for surgery will receive the preoperative 68Ga-MY6349 PET/CT in addition to standard MRI. Tumor uptake is quantified by the maximum standardized uptake value (SUVmax). The diagnostic performance of 68Ga-MY6349 PET is subsequently compared with MRI and the SUVmax is correlated with Trop2 expression levels in postoperative pathological specimens.

ELIGIBILITY:
Inclusion criteria:

* must be able to provide a written informed consent
* radiologically presumed and/or histologically confirmed craniopharyngioma scheduled for resection
* adequate clinical condition (Karnofsky performance status ≥70)

Exclusion criteria:

* concomitant major central nervous system disorders
* severe hepatic or renal dysfunction
* history of severe allergy or hypersensitivity to intravenous radiographic contrast agents
* claustrophobia precluding PET/CT or MRI examinations
* pregnancy or breastfeeding

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-MY6349 in PET imaging of craniopharyngioma | Within 1 week after PET imaging.
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in craniopharyngioma will be measured.

SECONDARY OUTCOMES:
Evaluate the feasibility of PET/CT imaging with 68Ga-MY6349 for the non-invasive assessment of Trop2 expression in craniopharyngioma. | Within 2 week after surgery.
  Trop2 expression analysis in tumor sample will be correlated to 68Ga-MY6349 tumor uptake, evaluated by measuring standardized uptake value (SUV) on the 68Ga-MY6349 PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Deling Li, MD, Study Chair — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China